CLINICAL TRIAL: NCT06484751
Title: Alberta Rehabilitation Advice Line SelfBack Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00142090
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The SelfBack app is a promising decision support system (DSS) App used globally to support and reinforce desired self-management behavior for LBP. Selfback's program goal is to improve the self-management of nonspecific LBP to reduce pain-related disability.
  Interventions: Device: SelfBack

INTERVENTIONS:
Device: SelfBack — The SelfBack app is a promising decision support system (DSS) App used globally to support and reinforce desired self-management behavior for LBP. Selfback's program goal is to improve the self-management of nonspecific LBP to reduce pain-related disability.

SUMMARY:
Recurrent and persistent low back pain (LBP) is a massive problem in Canada that causes a substantial pain, disability, cost, and even premature death.

The good news is that treatments for recurrent and persistent LBP are available. Many guidelines now recommend education and exercise as the best intervention for chronic LBP. Unfortunately, education and exercise programs are not publicly funded in Canada-only Canadians with extended health benefits can access these programs.

As a result, the 50% of Canadians who do not have extended health benefits often seek care for LBP from their publicly funded physicians. Physicians, in turn, have little choice but to reach for what they have available, including opioids, x-rays and referrals to specialists. Not only are these interventions unhelpful for chronic LBP, they are often harmful, sometimes deadly, and disproportionately affect lower socio-economic status households.

A possible solution to this problem exists in a validated app (SelfBack) that provides tailored self-management plans consisting of advice on physical activity, physical exercises, and educational content. Tailoring of treatment plans to individuals is achieved by using case-based reasoning methodology which is a branch of artificial intelligence.

This study will evaluate the feasibility of distributing the SelfBack app to persons experiencing LBP through the Rehabilitation Advice Line, a telephone service open Monday to Friday and provides rehabilitation advice and general health information for Albertans of any age.

The results of this study will help us understand the barriers and facilitators of distributing and using the app in the general pollution of Alberta. This information will be used to apply for funding for a larger study to understand the effectiveness of the app as an intervention for persistent and recurrent LBP.

DETAILED DESCRIPTION:
Purpose

This study will evaluate the feasibility of distributing the SelfBack app through the Rehab Avice Line and the feasibility of patients using the app.

Justification

The SelfBack app is a promising decision support system (DSS) App used globally to support and reinforce desired self-management behavior for LBP. Selfback's program goal is to improve the self-management of nonspecific LBP to reduce pain-related disability (Svenden, Sandal et al 2020). Using mHealth applications (apps) has been suggested to be a promising way to increase the effectiveness of self-management interventions (Beatty et al 2013, Newman et al 2011).

Objectives

Our primary objective is to evaluate the feasibility of distributing and using the SelfBack app. A secondary objective is to assess patient outcomes collected by the SelfBack app.

Methodology Overview

The Rehabilitation Advice Line will train their employees in the use of the SelfBack and how to distribute this app to patients. Rehab Advice Line employees are either licensed physiotherapists or occupational therapists. Those patients will be those Albertans who call the Rehab Advice Line and have a complaint of chronic low back pain (cLBP). Patients who are eligible and consent to participate will be provided with the SelfBack App. The SelfBack app then collects patients' data and provides patients with personalized advice regarding education and exercise for cLBP. De-identified group-level Selfback data will then be downloaded by the investigative team at regular intervals for analysis.

Overall timeline and setting:

The study will occur between May 2024 to December 2024 (8 months).

Recruitment and Inclusion/ Exclusion criteria:

Patient Recruitment: Rehab Advice Line Employees will identify potential patients through encounters with Albertans who call into the service. They will then discuss the study with those patients. Interested patients and those meeting the inclusion/exclusion criteria will be instructed on how to download the SelfBack app for use on their smartphone. They will then be sent an electronic information/consent form (via REDCap) by the Rehab Advice Line clinician. The phone call will then end. following the phone call, if the potential participant provides consent, the investigative team will be notified via REDCap and will then provide an activation code to the participant to activate the SelfBack app.

Patient Inclusion Criteria: Patients with persistent and/or recurrent LBP. Those who benefit most from Selfback are those who have persistent pain when defined as those currently having LBP that has impacted daily activities for > 1 month. In addition, eligible patients will...

be Albertan adults over 18 years of age be persons who meet the above definition of LBP, but may also include patients with stable radiculopathy/sciatica have a personal smartphone with internet access. have a working e-mail address. speak, read, and write English or have regular access to persons who can assist in this regard.

Ineligible patients will:

be patients who have complex back pain that requires direct clinical oversight. have cognitive impairments or learning disabilities limiting participation. have a serious mental illness have non-LBP illnesses or conditions that are contraindicated to participation in SelfBack (e.g. exercise).

have a terminal illness have an inability to take part in exercise/physical activity. Patient Data

Once the app is activated on the participant's smartphone, the SelfBack app will ask a series of baseline questions (~ 30 min) to establish what educational advice and exercises best suit the participant.

The SelfBack app regularly asks questions of the user to determine their ability to participate in exercise and education and evaluate their progress in the program. The list of survey questions used by the app was created, approved, and distributed by Selfback and is attached to this protocol.

The SelfBack will collect two categories of data.

The first category will be related to patient demographics.

The second category is related to patient-related outcome measures, a variety of established scales, and questionnaires with known psychometric properties. These outcome measures are used to assess the participant's health status, fitness level, and psychological health. These specific outcomes are asked at baseline, 3, and 6 months. A list of the patient-reported outcome measures used by SelfBack follows.

Roland-Morris Disability Questionnaire (RMDQ): The RMDQ is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. The RMDQ has been shown to yield reliable measurements, which are valid for inferring the level of disability, and to be sensitive to change over time for groups of patients with low back pain.

The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. The PSEQ is a useful tool for assessing an individual's self-efficacy beliefs related to pain management and for identifying individuals who may benefit from interventions to improve their pain management skills and self-efficacy.

EuroQol (EQ5D). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analog scale where the endpoints are labeled 'The best health you can image' and 'The worst health you can image (0-100). The VAS can be used as a quantitative measure of health outcomes that reflects the patient's judgment.

STarT Back: A simple tool to match patients to treatment packages appropriate for them. It has been shown to: significantly decrease disability from back pain, reduce time off work, and save money by making better use of health resources. This questionnaire helps clinicians identify modifiable risk factors (biomedical, psychological, and social) for back pain disability. The resulting score can stratify patients into low, medium, or high-risk categories. This tool can also be used to track change over time.

Numeric Pain Rating Scale (NPRS): A 0-10 NPRS ('0' no pain, and "10" worst pain imaginable) will be used to assess LBP intensity. The NPRS has excellent test-retest reliability. Previous research has found the NPRS to be responsive to change, with an MCID of 2 points for patients with acute LBP.

Psychosocial Covariate Measures: The Fear-Avoidance Beliefs Questionnaire (FABQ) will be used to measure patients' beliefs about how physical activity and work may affect their LBP and perceived risk for re-injury. The FABQ work score is a factor in the clinical prediction rule.

Clinician - Patient Interaction

Rehab Advice Line staff are also provided with a real-time dashboard where they can receive information about SelfBack users in real-time. Specifically, the dashboard shows if triggers have occurred that indicates the patient has entered information into the app that requires monitoring or follow-up (e.g. a sudden increase in pain).

Analyses

The general procedure for statistical analysis is as follows:

Descriptive statistics will be generated which will be cross-tabulated with demographic groups of interest (e.g., gender, age, community size, caregiver status, self-identification of disability, and ethnic and racial identification).

Feasibility will be judged as successful if 50% of the enrolled participants complete the education and exercise program recommended by the app.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria: Patients with persistent and/or recurrent LBP. Those who benefit most from Selfback are those who have persistent pain when defined as those currently having LBP that has impacted daily activities for > 1 month. In addition, eligible patients will...

* be Albertan adults over 18 years of age
* be persons who meet the above definition of LBP, but may also include patients with stable radiculopathy/sciatica
* have a personal smartphone with internet access.
* have a working e-mail address.
* speak, read, and write English or have regular access to persons who can assist in this regard.

Exclusion Criteria:

* be patients who have complex back pain that requires direct clinical oversight.
* have cognitive impairments or learning disabilities limiting participation.
* have a serious mental illness
* have non-LBP illnesses or conditions that are contraindicated to participation in SelfBack (e.g. exercise).
* have a terminal illness
* have an inability to take part in exercise/physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who utilize the SelfBack app | 12 months
  Success will be defined as 50% of patients using the app

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta rehabilitation advice line, Edmonton, Albertta, Canada

IPD SHARING:
Plan to Share IPD: No